CLINICAL TRIAL: NCT03843879
Title: A Comparison of Transversus Abdominis Plane Blocks Versus Continuous Intravenous Lidocaine for Kidney Transplant Surgery
Brief Title: TAP Blocks vs. IV Lidocaine for Kidney Transplants
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benaroya Research Institute (Other)
Responsible Party: Principal Investigator, Neil Hanson, Anesthesiologist, Benaroya Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB18-109
Record Dates: First submitted 2019-02-14; First posted 2019-02-18 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- TAP Block (Active Comparator): Single-injection transversus abdominis plane block
  Interventions: Procedure: Transversus Abdominis Plane Block
- IV Lidocaine (Active Comparator): Continuous intravenous lidocaine infusion
  Interventions: Drug: Intravenous Lidocaine

INTERVENTIONS:
Procedure: Transversus Abdominis Plane Block — Single-injection transversus abdominis plane block with 30 mL of 0.25% Bupivacaine with 1:400,000 epinephrine
  Other Names: TAP Block
  Arms: TAP Block
Drug: Intravenous Lidocaine — Continuous intravenous lidocaine infusion
  Other Names: Continuous intravenous lidocaine
  Arms: IV Lidocaine

SUMMARY:
This study will compare continuous intravenous lidocaine against single-injection transversus abdominis plane (TAP) block as a modality for postoperative analgesia in kidney transplant surgery.

DETAILED DESCRIPTION:
This study is a non-inferiority trial designed to assess the analgesic efficacy of an intravenous (IV) lidocaine infusion against single-injection transversus abdominis plane (TAP) block in patients undergoing kidney transplant surgery. The investigators propose a study of 124 subjects randomized into two groups. The control group will receive a TAP block. The study group will receive a continuous IV lidocaine infusion. The investigators hypothesize that there will be no statistically significant difference in postoperative opioid consumption between the two groups in the first 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipient
* >18 years old
* Consent to participate

Exclusion Criteria:

* <18 years old
* Refusal to participate
* Chronic opioid use
* Seizure disorder
* Allergy to local anesthestics
* Severe hepatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Opioid Consumption | 0-24 Hours
  Total opioid utilization

SECONDARY OUTCOMES:
Pain Scores | 0-48 Hours
  Numerical Rating Scale Pain Scores (Range: 0-10, where 0 is no pain and 10 is the worst pain)
Opioid Consumption | 24-48 Hours
  Total opioid utilization
Opioid-Related Adverse Events | 0-48 Hours
  Nausea, Vomiting, Pruritis, Respiratory Depression, Constipation
Block/Infusion-Related Adverse Events | 0-48 Hours
  Local Anesthetic Systemic Toxicity
Opioid Usage | 30 days from discharge
  Use of prescribed opioids

CONTACTS AND LOCATIONS:
Overall Officials: Neil A Hanson, MD, Principal Investigator — Virginia Mason Medical Center
Locations (1):
- Virginia Mason Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hanson NA, Strunk J, Saunders G, Cowan NG, Brandenberger J, Kuhr CS, Oryhan C, Warren DT, Slee AE, Strodtbeck W. Comparison of continuous intravenous lidocaine versus transversus abdominis plane block for kidney transplant surgery: a randomized, non-inferiority trial. Reg Anesth Pain Med. 2021 Nov;46(11):955-959. doi: 10.1136/rapm-2021-102973. Epub 2021 Aug 20. PMID 34417343